CLINICAL TRIAL: NCT06416618
Title: Surgical Versus Non-surgical Treatment of Displaced Proximal Humerus Fracture in Adults Aged 50 to 65 Years: a Pragmatic Randomized Controlled Trial
Brief Title: Surgical Versus Non-surgical Treatment of Displaced Proximal Humerus Fracture in Adults Aged 50 to 65 Years
Acronym: PHF50-65
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Line Lojbert Houkjaer, Principal Investigator, M.D., Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHF5065
Record Dates: First submitted 2024-05-08; First posted 2024-05-16 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Proximal Humeral Fracture; Shoulder Fractures
MeSH Terms: conditions — Shoulder Fractures | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: The study is a two-center, parallel-group, randomized, superiority trial
Who Masked: Outcomes Assessor
Masking Description: The primary investigator will conduct the blinded statistical analysis through data anonymization and will be supervised by a biostatistician. After the blinded statistical analysis has been completed, two abstracts will be written based on the pre-blinding analysis results before the blinding is revealed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-surgical treatment (Experimental): Patients in the non-surgical group will be offered an optional sling for comfort for an additional 1-2 weeks at their first visit,
  Interventions: Procedure: Non surgical
- Procedure: Surgical treatment (Active Comparator): The surgical group will receive osteosynthesis with a locking plate or an intramedullary locking nail, according to the surgeon's choice
  Interventions: Procedure: Surgical

INTERVENTIONS:
Procedure: Surgical — Surgical group: After osteosynthesis, they will be provided with a sling and swathe immediately after the surgery. From the first postoperative day, only the sling will be used. Two weeks postoperatively, patients will undergo clinical and radiological follow-up in the outpatient clinic. They will be referred to post-operative rehabilitation in the municipalities. At 12 weeks postoperatively, patients will have another clinical and radiological follow-up. This is the current standard care for surgical treatment with a plate or intramedullary nail.
  Arms: Procedure: Surgical treatment
Procedure: Non surgical — Non-surgical group: Patients in the non-surgical group will be offered an optional sling for comfort for an additional 1-2 weeks at their first visit, 10-14 days post-injury. Patients will be referred to rehabilitation in the municipalities. At week 6 post-injury, all patients will undergo clinical and radiological follow-up. This represents the current standard care for non-surgical treatment of displaced PHF at the departments.
  Arms: Non-surgical treatment

SUMMARY:
The goal of this clinical trial is to study whether surgery results in better functional outcomes than non-surgical treatment among patients aged 50-65 with a displaced proximal humerus fracture.

The main questions it aims to answer are:

• Does osteosynthesis result in better patient-reported functional outcomes compared to non-surgical treatment at 12 months follow-up?

Aim is also to characterize the patient group aged 50-65 regarding fracture morphology, osteoporosis, and clinical frailty scale.

The study compare operation with either plate or nail fixation to non-surgical treatment.

Participants will:

* Receive either surgical treatment or non-surgical treatment.
* At 6 months, 1 year, and 2 years, the patient will answer two short questionnaires (Oxford Shoulder Score and Eq-5D-3L).

The primary outcome will be Oxford Shoulder Score at 12 months. The secondary outcome will be OSS at 6 and 24 months and EQ-5D-3L score measured at the same time-points. Adverse events and conversion to surgery will be registered. OSS and EQ-5D-3L will be completed just before the 6 months visit.

DETAILED DESCRIPTION:
Proximal humerus fractures (PHF) are common injuries. At the age of 60 and above, no clinically important difference between surgical and non-surgical treatment after one year has been reported based on a recent Cochrane review of 10 trials.

The treatment of choice for displaced PHF in adults 50-65 years is anatomical reconstruction, and osteosynthesis if possible, which is why many patients in this age group with a displaced PHF undergo surgical treatment.

Orthopaedic surgeons may encounter challenges in guiding patients and formulating treatment strategies within specific age groups due to the absence of inclusion of this younger patient demographic in existing evidence. Knowledge is primarily derived from studies on the population aged 60 years and above. There exists an intermediate age group of patients for whom it remains uncertain whether the benefits and harms of non-surgical and surgical interventions are comparable

This trial is a two-center, parallel-group, randomized, superiority trial comparing osteosynthesis with non-surgical treatment following a displaced proximal humerus fractures in patients aged 50-65 years. The participants will be included and allocated equally to surgical treatment with osteosynthesis (comparator) with non-surgical treatment (intervention).

The surgical group will visit the outpatient clinic after 2, 12, and 24 weeks, while the non-surgical group will visit after 6, (12) and 24 weeks. X-rays will be obtained before every visit.

Both groups will be referred to rehabilitation in the municipalities.

Without a patient-derived MCID for PHF, a relevant difference of 9,6 was assumed to represent clinically meaningful difference. This is equivalent to approximately a 20 % difference between the surgical group and the non-surgical group on a 0-48 OSS scale. With a power of 80% and a 5% level of significance, a sample size of 25 participants per group is required. Assuming a 15 % loss to follow-up, the recruitment target is 30 patients in each group, meaning 60 participants overall.

In case of treatment failure in either group, defined as persistent pain or a failed osteosynthesis, a salvage procedure with secondary osteosynthesis or a reverse shoulder arthroplasty (RSA), will be offered.

Additionally, there are plans for a systematic collection of reasons for non-inclusion of eligible patients who were not recruited into the trial (decliner cohort), and their baseline characteristics, treatment preferences. The decliner cohort will receive the same treatment, follow-up, and outcome measurements as the included patients.

Statistical analysis:

Baseline characteristics will be presented using descriptive statistics. Investigators will compare the following patient characteristics between the groups at baseline: age (categorized into 5-year age groups), sex, height, weight, ASA score, fracture classification (Neer), dominant arm (yes/no), smoking, alcohol consumption, educational level, working status, work type, osteoporosis (three-level ordinal variable based on T-scores (osteoporosis, osteopenia, and normal bone density)) and clinical frailty scale. SD will be reported, and n (%) for categorical values.

Osteoporosis will be collected and reported descriptively as a three-level ordinal variable based on T-scores (osteoporosis, osteopenia, and normal bone density).

The OSS results for surgical and non-surgical treatment groups at 6, 12, and 24 months will be tabulated and graphically represented with mean, SD, median, and IQR according to the distribution.

The primary outcome, OSS at 12 months, will be analysed using two-sample t-test comparing the two treatment groups. Normality assumptions will be assessed, and if violated, alternative methods such as transformation or non-parametric Mann-Whitney U test will be considered. As suggested in the extension of the CONSORT 2010 statement, the primary outcome will be analysed for the intention-to-treat (ITT) population.

In addition, linear mixed models will be used to analyse OSS and EQ-5D over time (6, 12 and 24 months) accounting for the repeated measures structure and to explore outcome trajectories. Model-based contrasts from the LMM will be used to estimate adjusted between-group differences at specific time points. Missing data will be handled within the mixed model framework, assuming data are missing at random. Details are provided in Supplementary Information, file 4.

Investigators will record and report adverse events in each group. At the 6-month follow-up, patients will be asked, and investigators will record and report the length of rehabilitation in municipalities (in weeks) and whether the patient has followed the rehabilitation plan.

Salvage procedure Salvage procedures and adverse events will be reported descriptively. Reoperation in the form of hardware removal will be classified as a complication, not a salvage procedure. There will be two analyses for ITT: one including salvage procedures and one excluding them. The timing of salvage procedures will be analyzed using a Cox proportional hazards model to compare time to salvage between treatment groups.

Non-randomized cohort (decliner cohort) Patients who declined randomization but consented to follow-up will form the non-randomized cohort. Baseline characteristics will be summarized descriptively and compared between the randomized and non-randomized cohorts, as well as among the non-randomized patients by treatment choice. The primary outcome (OSS at 12 months) will be analyzed by treatment modality. Secondary outcome measures (OSS and EQ-5D) will be presented descriptively and graphically at 6, 12, and 24 months. Analyses will include multivariable linear regression adjusted for baseline covariates; propensity score methods may be applied. The incidence and timing of salvage procedures will be described and analyzed using Cox proportional hazards models.

Blinded data interpretation Although patients and investigators are not blinded to treatment allocation, the primary investigator will conduct blinded statistical analysis through data anonymization and will be supervised by a biostatistician. The OSS and EQ-5D-3L will be completed just before the 6-month visit, collected automatically through REDCap, and will not be reviewed by the investigator prior to analysis- After the blinded statistical analysis has been completed, two abstracts will be written based on the pre-blinding analysis results before the blinding is revealed.

Data will be analysed using the statistical "R" .

Interim analyses An interim analysis will be conducted when 50% (n = 30) of the randomized patients have completed their 6-month follow-up, focusing on OSS, failure to treatment, and serious complications. A third party will blind the data to treatment location before analysis. Regardless of whether the interim analyses suggest that the study is unlikely to achieve its primary objectives, the study will proceed as initially planned.

A DMC has been organized to monitor and evaluate the data from the interim analysis. The DMC consists of four independent members, including four orthopedic researchers and an orthopedic nurse.

The DMC will monitor unexpected, unwanted events; continued inclusion will be considered if the failure rate is above 30 %. Intervention-related hospitalization or mortality will be reported to the ethics committee.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 50 and 65 years with a displaced PHF assessed to be constructible by the treating surgeon after a low-energy trauma will be considered for eligibility.
* Patients should be cognitively capable of answering the follow-up questionnaires.

Exclusion Criteria:

* The patient does not understand written and spoken native language (Danish or Finnish/Swedish)
* Inability to give informed consent
* Fractures assessed to be unreconstructedly by the treating surgeon
* Isolated tuberosity fracture, fracture dislocations, open fractures, and fractures with involvement of the articular surface
* Less than 25% contact between head fragment and metaphysis/diaphysis measured at two perpendicular radiographs at two weeks.
* Pathological fractures or previous fractures in the same proximal humerus
* Concomitant fractures, which could influence the outcome
* Paralysis in upper extremity

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Oxford Shoulder Score 12 months | 12 months
  Oxford Shoulder Score is a patient-reported shoulder-specific outcome measure. It is a patient-administrated questionnaire to assess shoulder function. It consists of 12 questions on a 5-point Likert scale (both pain- and function-related), each offering five ordinal response options. The cumulative score ranges between 0 and 48, being 0 (worst) to 48 (best: no pain or no functional limitation).

SECONDARY OUTCOMES:
Oxford Shoulder Score | 6 and 24 months
  Oxford Shoulder Score is a patient-reported shoulder-specific outcome measure. It is a patient-administrated questionnaire to assess shoulder function. It consists of 12 questions on a 5-point Likert scale (both pain- and function-related), each offering five ordinal response options. The cumulative score ranges between 0 and 48, being 0 (worst) to 48 (best: no pain or no functional limitation).
EQ-5D-3L | 6, 12 and 24 months
  Q-5D-3L is a generic health-related quality-of-life assessment tool. It consists of a 5-dimension descriptive questionnaire about mobility, self-care, usual activities, pain/discomfort, and anxiety/depression as a measure for health-related quality of life. Each dimension has 3 levels: No problems, some/moderate problems and unable/extreme problems. Each dimension is weighted differently and results in a total score based on the EQ-5D index calculator (TTO). The EQ-5D-3L also includes an overall scale (numeric rating scale) in which patient rates overall health condition today on a scale between 1 - 100, with 100 being the highest level of health imaginable
Conversion to surgery after inclusion, or additional surgery | 24 months
  Treatment failure: In case of treatment failure in either group, defined as persistent pain or a failed osteosynthesis, a salvage procedure with secondary osteosynthesis, including the possibility to use graft or a reverse shoulder arthroplasty (RSA), will be offered. Failed osteosynthesis and the most appropriate salvage procedure will be defined by the surgeon.
  Cross-over to reverse shoulder arthroplasty or revision osteosynthesis is considered a failure of treatment regardless of group allocation. The patient will remain in the study. The reason for crossing over will be noted and reported.
Adverse events. | 24 months
  Serious adverse events, as defined by the WHO. Systemic reviews on terms and definitions for complications after surgical and non-surgical treatment have been conducted. Based on international consensus on the core event set for PHF, both surgical and non-surgical treatment, 8 event groups are defined. The following adverse event groups will be monitored: implant, osteochondral, shoulder instability, peripheral neurology, vascular, infection, device, superficial soft tissue, and deep soft tissue. In addition to this, we have chosen to monitor clinical symptoms such as persistent severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Line Løjbert Houkjær, M.D., Principal Investigator — Center for evidensbaseret ortopædkirurgi, Sjællands Universitets Hospital, Køge.
Locations (2):
- Centre for Evidence-Based Orthopaedics, Zealand University Hospital, Køge, Region Sjælland, Denmark
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196
- [Background] Alispahic N, Brorson S, Bahrs C, Joeris A, Steinitz A, Audige L. Complications after surgical management of proximal humeral fractures: a systematic review of event terms and definitions. BMC Musculoskelet Disord. 2020 May 26;21(1):327. doi: 10.1186/s12891-020-03353-8. PMID 32456631
- [Background] Brorson S, Alispahic N, Bahrs C, Joeris A, Steinitz A, Audige L. Complications after non-surgical management of proximal humeral fractures: a systematic review of terms and definitions. BMC Musculoskelet Disord. 2019 Feb 23;20(1):91. doi: 10.1186/s12891-019-2459-6. PMID 30797232
- [Background] Audige L, Brorson S, Durchholz H, Lambert S, Moro F, Joeris A. Core set of unfavorable events of proximal humerus fracture treatment defined by an international Delphi consensus process. BMC Musculoskelet Disord. 2021 Nov 30;22(1):1002. doi: 10.1186/s12891-021-04887-1. PMID 34847888
- [Derived] Houkjaer L, Launonen AP, Sumrein BO, Karna L, Issa Z, Holtz KB, Brorson S. Surgical versus non-surgical treatment of proximal humerus fracture in patients aged 50-65 years: young shoulder CARE (displaCed proximAl humeRus fracturE) trial-a pragmatic randomized controlled trial study protocol. Trials. 2025 Dec 29;26(1):588. doi: 10.1186/s13063-025-09283-x. PMID 41466383
- See also: EMEA: Clinical Safety Data Management: Definitions and Standards for Expedited Reporting — https://www.ema.europa.eu/en/documents/scientific-guideline/international-conference-harmonisation-technical-requirements-registration-pharmaceuticals-human-use-topic-e-2-clinical-safety-data-management-definitions-and-standards-expedited-reporting-step_en.pdf